CLINICAL TRIAL: NCT05548322
Title: Studies Into Touch in Healthy Humans to Provide Sensory Feedback in Prostheses
Acronym: TACTHUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C21-19; 2021-A01604-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-09-02; First posted 2022-09-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Somatosensory Disorders; Amputation; Tactile Disorders; Aging; Prosthesis User
Keywords: Touch; Temperature; Somarosensation; Prosthetics; Microneurography; Tactile; Mechanoreceptor
MeSH Terms: conditions — Somatosensory Disorders | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will take part in experiments that investigate the seven arms of the study. Participants with an amputation will only take part in arm 7. Healthy participants may take part in one to six arms (arms 1-6). However, this is dependent upon the recordings found in the experiment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Study of tactile afferent responses to natural surfaces (Experimental)
  Interventions: Device: Different surfaces to be touched
- Modulation of touch according to the emotional state (Experimental)
  Interventions: Device: Different surfaces to be touched; Behavioral: Emotional state change
- Effect of temperature on tactile sensitivity (Experimental)
  Interventions: Device: Different surfaces to be touched
- Origin of wetness perception (Experimental)
  Interventions: Device: Different surfaces to be touched
- Aging and tactile sensitivity (Experimental)
  Interventions: Device: Different surfaces to be touched; Behavioral: Emotional state change; Device: Electrical stimulation
- Tactile perceptions induced by the stimulation of single sensory fibers (Experimental)
  Interventions: Device: Electrical stimulation
- Study of tactile feedback after amputation (Experimental)
  Interventions: Device: Different surfaces to be touched; Device: Electrical stimulation

INTERVENTIONS:
Device: Different surfaces to be touched — The participant will touch various different surfaces and textures, including ones of different temperature and including solids and liquids.
  Arms: Aging and tactile sensitivity; Effect of temperature on tactile sensitivity; Modulation of touch according to the emotional state; Origin of wetness perception; Study of tactile afferent responses to natural surfaces; Study of tactile feedback after amputation
Behavioral: Emotional state change — The emotional state of the participant will be modulated by listening to music.
  Arms: Aging and tactile sensitivity; Modulation of touch according to the emotional state
Device: Electrical stimulation — The participant will receive electrical stimulation of single nerve fibers (a few microamps) to artificially excite an individual afferent.
  Arms: Aging and tactile sensitivity; Study of tactile feedback after amputation; Tactile perceptions induced by the stimulation of single sensory fibers

SUMMARY:
Our sense of touch is essential to explore our environment and experience life and is based on signals from receptors in the body that are sensitive to different types of stimulation. The TACTHUM projects aims to investigate the fundamental firing of mechanoreceptors in the body to various external stimuli, with an end-aim to better understand the human somatosensory system and to apply this knowledge to provide comprehensive sensory feedback in prosthetics. We have a vast system of peripheral receptors in the skin and muscles that provide us with exquisitely detailed information about our everyday interactions. When there is injury to a body part, such as in amputation, there is a significant loss of somatosensory input. Prosthetic devices have greatly developmed in the past few years, especially with the introduction of useful sensory feedback. However, there is a lot to discover both about the workings of the somatosensory system and how to recreate this to give feedback in a prosthetic device.

The main objective of the TACTHUM project is to understand how to recover and apply useful somatosensory feedback in prostheses for amputees. There are a number of other sub-objectives, to:

1. Determine how tactile mechanoreceptors encode the texture of natural surfaces during passive and active exploration.
2. Investigate how our sense of touch varies with emotional state.
3. Explore what happens to our sense of touch when we explore surfaces at different temperatures.
4. Understand the origin of our perception of humidity.
5. Investigate differences in the encoding of tactile information with age.
6. Determine the perceptions generated by the stimulation of single tactile afferents.
7. Study changes in spontaneous activity and responses to tactile stimulation on the residual limb of amputees.

To accomplish these objectives, we will primarily use the technique of microneurography, in vivo recordings from peripheral nerves, to gain direct information about the firing of peripheral neurons in humans. In conjunction with this, we will use a variety of mechanical and thermal stimuli to excite somatosensory fibers and register the activity of other physiological and perceptual measures. This will allow us to gain a fuller understanding of how the incoming somatosensory signals are interpreted and processed. Overall, we aim to explore how more naturalistic tactile interactions are encoded and how these can be translated to provide realistic prosthetic feedback.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 70.
* Be a member of a social security scheme, or a beneficiary of such a scheme
* Be calm enough to sit still for four hours.
* Specific for people participating in Arm 7 on amputees: People with an upper or lower limb amputation (unilateral) of more than 2 years.

Exclusion Criteria:

* Have peripheral neuropathy (diabetes, Raynaud's disease) or chronic muscle and/or sensory pain.
* Have a neurological or psychiatric history.
* Be subject to epilepsy.
* Be pregnant (declared) or breastfeeding, having given birth within the last year.
* Be afraid of injections.
* Being under dermatological treatment.
* Have a pacemaker.
* Not being able to understand the information leaflet and the consent form or sign it.
* Be subject to a legal protection measure (declarative)
* Be a protected adult (curatorship or guardianship)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2034-10-02 (Estimated); Study Completion 2034-11-02 (Estimated)

PRIMARY OUTCOMES:
Microneurography recording | Measured during the experiment (single event, max. 6 hours), during stimulation intervention
  The discharge of a peripheral nerve fiber will be recorded during the stimulation conditions. From this recording, measures of the total number of impulses evoked, the instantaneous and average frequencies, firing variability, and frequency composition will be extracted.

SECONDARY OUTCOMES:
Electrodermal response | Measured during the experiment (single event, max. 6 hours), during stimulation intervention
  Electrodermal response will be recorded from electrodes attached to the glabrous skin, to register further effects of the stimulation on the body.
Heart rate | Measured during the experiment (single event, max. 6 hours), during stimulation intervention
  Heart rate will be recorded via three electrodes on the skin, to register further effects of the stimulation on the body.
Electromyography | Measured during the experiment (single event, max. 6 hours), during stimulation intervention
  Electromyography (EMG) will be recorded from surface skin electrodes over the muscle, to register further effects of the stimulation on the body. From this recording, measures of the total activity (area under the curve) during a stimulation period and the frequency composition will be extracted.
Electroencephalography | Measured during the experiment (single event, max. 6 hours), during stimulation intervention
  Electroencephalography (EEG) will be recorded from surface scalp skin using a 64 electrodes setup, to register further effects of the stimulation on brain responses. From this recording, measures of the event-related potentials to stimulation will be analyzed and the frequency composition (theta, alpha, beta, gamma) of the response will be extracted.
Perceptual ratings of pleasantness | Measured during the experiment (single event, max. 6 hours), directly after the stimulation intervention
  The perceptual rating of the perceived pleasantness of different applied stimuli will be gained to determine the overt sensations induced by the stimulation. The scale is a visual analog scale with the anchors 'pleasant' and 'unpleasant' that outputs a scale of 0 (unpleasant) to 100 (pleasant).
Perceptual ratings of roughness | Measured during the experiment (single event, max. 6 hours), directly after the stimulation intervention
  The perceptual rating of the perceived roughness of different applied stimuli will be gained to determine the overt sensations induced by the stimulation. The scale is a visual analog scale with the anchors 'smooth' and 'rough' that outputs a scale of 0 (smooth) to 100 (rough).
Perceptual ratings of intensity | Measured during the experiment (single event, max. 6 hours), directly after the stimulation intervention
  The perceptual rating of the perceived intensity of different applied stimuli will be gained to determine the overt sensations induced by the stimulation. The scale is a visual analog scale with the anchors 'not al all intense' and 'intense' that outputs a scale of 0 (not at all intense) to 100 (intense).

CONTACTS AND LOCATIONS:
Overall Officials: Maya Elzeiere, MD, Principal Investigator — CNRS - Aix-Marseille University; Rochelle Ackerley, PhD, Study Director — CNRS - Aix-Marseille University
Locations (2):
- France (2):
  - CNRS - Aix-Marseille University UMR7291, Marseille
  - Hôpital HIA Lavéran, Marseille

IPD SHARING:
Plan to Share IPD: Undecided